CLINICAL TRIAL: NCT01809769
Title: Autologous Adipose Tissue Derived Mesenchymal Stem Cells Therapy for Patients With Knee Osteoarthritis by Intra-articular Injection: A PhaseⅠ/Ⅱa, Randomized and Double-blinded Clinical Trial
Brief Title: Autologous Adipose Tissue Derived Mesenchymal Stem Cells Therapy for Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CBMG-KOA-1.1
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mesenchymal stem cells low-dose group (Experimental): Biological: Mesenchymal progenitor cells. Administrated for intra-articular use. Dosage: 1 x 10 E7 cells (3 ml), Frequency: 0,3 weeks.
  Interventions: Biological: Mesenchymal stem cells low-dose group
- Mesenchymal stem cells mid-dose group (Experimental): Biological: Mesenchymal progenitor cells. Administrated for intra-articular use. Dosage: 2 x 10 E7 cells (3 ml). Frequency: 0,3 weeks.
  Interventions: Biological: Mesenchymal stem cells mid-dose group
- Mesenchymal stem cells high-dose group (Experimental): Biological: Mesenchymal progenitor cells. Administrated for intra-articular use. Dosage:5 x 10 E7 cells (3 ml). Frequency: 0,3 weeks.
  Interventions: Biological: Mesenchymal stem cells high-dose group

INTERVENTIONS:
Biological: Mesenchymal stem cells low-dose group — Biological: Adipose tissue derived mesenchymal stem cells administrated for intra-articular use
  Other Names: Adipose tissue derived mesenchymal stem cells
  Arms: Mesenchymal stem cells low-dose group
Biological: Mesenchymal stem cells mid-dose group — Biological: Adipose tissue derived mesenchymal stem cells administrated for intra-articular use
  Other Names: Adipose tissue derived mesenchymal stem cells
  Arms: Mesenchymal stem cells mid-dose group
Biological: Mesenchymal stem cells high-dose group — Biological: Adipose tissue derived mesenchymal stem cells administrated for intra-articular use
  Other Names: Adipose tissue derived mesenchymal stem cells
  Arms: Mesenchymal stem cells high-dose group

SUMMARY:
Two injections in total and 3 ml autologous adipose-tissue-derived stem cells(haMSCs) for each injection; time-points for intervention: 1) initial injection; 2) 3 weeks following initial injection.

DETAILED DESCRIPTION:
Adipose (fat) tissue is removed by lipo-aspiration (this may take up to 40 minutes). The fat is processed on-site to isolate and obtain the MSCs,then proliferate them. The suspension of the cells is injected into the knee joint under ultrasound guidance. (about 20 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and sign the consent form for this study.
* Age: 40-70, males and females.
* Clinical diagnosis of degenerative arthritis by Radiographic Criteria of Kellgren and Lawrence.
* Patients who can't treat with traditional medication and need a arthroplasty.
* Duration of pain over Grade 4(11-point numeric scale)> 4 months.

Exclusion Criteria:

* Women who are pregnant or breast feeding or planning to become pregnant during the study.
* Objects who administer with a anti-inflammatory drugs within 14 days prior to inclusion in the study.
* History or current evidence of alcohol or drug abuse or is a recreational user of illicit drugs or prescription medications.
* Treatment with intra-articular injection therapy within 2 months prior to screen.
* Other joint diseases except degenerative arthritis : systemic or rheumatic or inflammatory chondropathy, chondrocalcinosis, hemachromatosis, inflammatory joint disease, avascular necrosis of the femoral head, Paget's disease, hemophilic arthropathy, infectional arthritis, Charcot's disease, villonodular synovitis, synovial chondromatosis.
* Positive serology for HIV-1 or HIV-2, Hepatitis B (HBsAg, Anti-HCV-Ab), Hepatitis C (Anti-HCV-Ab) and syphilis.
* Serious pre-existing medical conditions like Cardiovascular Diseases, Renal Diseases, Liver Diseases, Endocrine Diseases, Cancer and Diabetes Mellitus.
* Overweight expressed as body mass index (BMI) greater than 30 (obesity grade II).
* Participation in another clinical trial or treatment with a different investigational product within 3 months prior to inclusion in the study.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Recording of Adverse Events and Serious Adverse Events | 12 weeks
Electrocardiogram | 9 weeks
Vital signs | 9 weeks
Physical examination | 9 weeks
WOMAC Score(The Western Ontario and McMaster Universities Osteoarthritis Index) | 24 months
Laboratory tests | 9 weeks
  Routine blood and urine tests, hepatic and renal functions tests, blood lipid and glucose tests, immunologic tests

SECONDARY OUTCOMES:
SF-36 | 24 months
NRS-11 | 24 months
The volume of articular cartilage | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, M.D. & Ph.D., Principal Investigator — Department of Rheumatology,Ren Ji Hospital,School of Medicine,Shanghai Jiao Tong University,Shanghai,China
Locations (1):
- Department of Rheumatology,Ren Ji Hospital,School of Medicine,Shanghai Jiao Tong University,Shanghai,China, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Song Y, Du H, Dai C, Zhang L, Li S, Hunter DJ, Lu L, Bao C. Human adipose-derived mesenchymal stem cells for osteoarthritis: a pilot study with long-term follow-up and repeated injections. Regen Med. 2018 Apr;13(3):295-307. doi: 10.2217/rme-2017-0152. Epub 2018 Feb 8. PMID 29417902